CLINICAL TRIAL: NCT05567549
Title: Frequency of Sarcopenia and Relation With Mortality in Elderly at the Emergency Department
Brief Title: Evaluation of Sarcopenia in Elderly at the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ozge Can. MD, MD, Ege University
Other Study IDs: 22-8.1T/60
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

SUMMARY:
The goal of this observational study is to evaluate in elderly patients for the frequency of sarcopenia and its relationship with mortality in a university hospital.

The main questions it aims to answer are;

1. What is the frequency of sarcopenia in elderly patients at emergency department?
2. Is sarcopenia associated with mortality in an elderly patient admitted to the emergency department?

ELIGIBILITY:
Inclusion Criteria:

1. Above the age of 65 admitted to the emergency department
2. Able to walk without support
3. No lower extremity fracture
4. No disease with neuromuscular involvement

Exclusion Criteria:

1. In the presence of a cerebrovascular event
2. Those in need of critical intervention when applying to the emergency department
3. Unconscious patients

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients over 65 years of age, who can walk independently, who do not have lower extremity fractures or neuromuscular disease, will constitute the study population.
  The mortality rate over the age of 65 was found to be 11%. Considering that the mortality rate with sarcopenia was 28%, it was found that 63 patients were required for the effect of sarcopenia on mortality with a 95% confidence interval and 0.5% margin of error. Since the incidence of sarcopenia in the emergency department was 33%, 200 patients were planned to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-10 (Estimated); Primary Completion 2023-07-10 (Estimated); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 0-28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morley JE. Sarcopenia: diagnosis and treatment. J Nutr Health Aging. 2008 Aug-Sep;12(7):452-6. doi: 10.1007/BF02982705. No abstract available. PMID 18615226
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Roberts S, Collins P, Rattray M. Identifying and Managing Malnutrition, Frailty and Sarcopenia in the Community: A Narrative Review. Nutrients. 2021 Jul 5;13(7):2316. doi: 10.3390/nu13072316. PMID 34371823
- [Background] Hung SK, Kou HW, Hsu KH, Wu CT, Lee CW, Leonard Goh ZN, Seak CK, Chen-Yeen Seak J, Liu YT, Seak CJ; SPOT investigators. Sarcopenia is a useful risk stratification tool to prognosticate splenic abscess patients in the emergency department. J Formos Med Assoc. 2021 Mar;120(3):997-1004. doi: 10.1016/j.jfma.2020.08.039. Epub 2020 Sep 9. PMID 32917483
- [Background] McQuade C, Kavanagh DO, O'Brien C, Hunter K, Nally D, Hickie C, Ward E, Torreggiani WC. CT-determined sarcopenia as a predictor of post-operative outcomes in patients undergoing an emergency laparotomy. Clin Imaging. 2021 Nov;79:273-277. doi: 10.1016/j.clinimag.2021.05.015. Epub 2021 May 18. PMID 34171595